CLINICAL TRIAL: NCT03567447
Title: Effect of L-Dihydroxyphenylserine (L-DOPS) on Falls in Patients With Neurogenic Orthostatic Hypotension (NOH)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: H. Lundbeck A/S (Industry); Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-0200-80-04
Record Dates: First submitted 2018-05-21; First posted 2018-06-25 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Parkinson Disease; Falls Patient
Keywords: Parkinsons Disease; PD; Patient Falls; Neurogenic Orthostatic Hypotension
MeSH Terms: conditions — Parkinson Disease | interventions — Droxidopa

STUDY DESIGN:
Intervention Model Description: Phase II single center, double-blind, randomized, placebo-controlled, efficacy study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): This group will receive droxidopa 100mg to 600mg three times a day (TID) titration for 2 weeks and then maintenance dosage for 4 additional weeks. We will assess participants two times over the 4-week intervention. Each assessment will be the same as the baseline assessment, including the Orthostatic Hypotension Symptom Assessment (OHSA), postural, and gait assessments, and will be administered during the 2nd and 4th weeks following onset of stable treatment phase.
  Interventions: Drug: Droxidopa; Other: Placebo
- Non treatment group (Placebo Comparator): This group will receive placebo appearing to be 100mg to 600mg three times a day (TID) titration for 2 weeks and then maintenance dosage for 4 additional weeks. We will assess participants two times over the 4-week intervention. Each assessment will be the same as the baseline assessment, including the Orthostatic Hypotension Symptom Assessment (OHSA), postural, and gait assessments, and will be administered during the 2nd and 4th weeks following onset of stable treatment phase.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Droxidopa — starting with 100 mg TID and increasing in 100 mg TID increments, to a maximum of 600mg TID, to identify the highest tolerated dose for each patient.
  Other Names: NORTHERA
  Arms: Treatment group
Other: Placebo — appearing to be 100 mg TID and increasing in 100 mg TID increments, to a maximum of 600mg TID, to identify the highest tolerated dose for each patient.

SUMMARY:
This will be a Phase II single center, double-blind, randomized, placebo-controlled, efficacy study. Subjects will complete six visits. The first will be a screening visit. There will be four assessment visits: baseline, 2 weeks after the double-blinded trial begins, the end of the blinded trial, and after 4 weeks of washout. There will also be an additional randomization and medication dispensing visit immediately following the dose optimization period and preceding the double-blinded trial.

DETAILED DESCRIPTION:
Injuries associated with falls continue to pose a significant burden to patients with Parkinson's disease (PD) both in terms of human suffering and economic losses. Overall annual fall incidence rates range from 50-70% for PD patients, and recurrent falls are a major cause of disability in PD. Approximately 20% of patients with Parkinson's disease develop NOH which can lead to falls. Although the mechanisms underlying impaired postural stability and falls are not well-known in patients with PD, attention is focused on the noradrenergic system. L-DOPS, a drug that enhances norepinephrine levels in peripheral and central nervous system, has been shown to moderate NOH, and often improve symptoms concomitant of PD and falls.

This study will help to determine the effect of L-DOPS in reducing falls and fall severity by using an instrumented walkway to induce slip perturbations can assess the propensity for falls and fall-related outcomes. It will assess fall events from the point of initiation through recovery. The effect of L-DOPS on gait and balance parameters will also be measured using force plate and inertial measurement unit (IMU) testing, and improvement in clinical scores such as the MDS-UPDRS will be monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has voluntarily signed and dated an informed consent form (ICF), approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), and provided Health Insurance Portability and Accountability Act (HIPAA) (or other applicable privacy regulation) authorization prior to any participation in the study.
2. Subject is male or female and is ≥ 30 and ≤ 83 years of age.
3. Parkinson's diagnosis with history of falls or gait difficulty.
4. Subject demonstrates neurogenic orthostatic hypotension (drop of 20 mm/Hg Systolic or 10 mm/Hg diastolic or both within 3 min of standing)
5. Fell more than once in past year.
6. Montreal Cognitive Assessment (MoCA) score ≥ 21.
7. Stable dose of levodopa, dopamine agonist, amantadine, and/or monoamine oxidase B inhibitor, i.e. unchanged for 1 month.
8. Subject is ambulatory and able to walk ≥ 10 meters with/without the use of an assistive device.

Exclusion Criteria:

1. Subject has a clinical diagnosis of an atypical Parkinsonism
2. Subject has a clinical diagnosis of PD that is suspicious to the investigator as being a possible case of atypical Parkinson's
3. History of significant psychiatric illness such as schizophrenia or bipolar affective disorder or any other significant psychiatric illness that in the opinion of the investigator would interfere with participation in the study; history of major depressive disorder in the past year, or current major depressive episode
4. Patients with systolic BP ≤70 mm/hg
5. Subjects with a history of coronary artery disease or congestive heart failure
6. Participation in another investigational drug or device study in during the 60 days prior to the Screening Visit
7. Treatment with any anti-hypertensive medications
8. Treatment with any anti-spasmodic medications
9. Treatment with medications intended to elevate blood pressure
10. Treatment with non-specific monoamine oxidase (MAO) inhibitors

Ages: 30 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-08-17 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in number of falls | Study weeks 2, 4 and 8
  The effect of L-DOPS on falls will be assessed by measuring the number of falls during balance perturbation testing.

SECONDARY OUTCOMES:
Change in objective and subjective measures of Balance | Study weeks 2, 4 and 8
  The effect of L-DOPS on assessments of balance by Movement Disorder Society- Unified Parkinson's Disease Rating Scale (MDS-UPDRS)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Lieberman, MD, Principal Investigator — Barrow Neurological Insitute
Locations (1):
- Barrow Neurological Institute at St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No